CLINICAL TRIAL: NCT04024657
Title: A Cross Sectional, Diagnostic Accuracy Study to Validate the Use of a New Device(Inflammacheck™) in Diagnosing COPD by Measuring the Level of Exhaled Breath Condensate Hydrogen Peroxide (EBC H2O2)
Brief Title: A Cross Sectional, Diagnostic Accuracy Study to Validate the Use of a New Device(Inflammacheck™) in Diagnosing COPD
Acronym: EXHALE 1V
Status: Completed | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: PHT/2018/71
Record Dates: First submitted 2019-05-03; First posted 2019-07-18 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: COPD Exacerbation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A cross-sectional, diagnostic accuracy study to evaluate the use of the 'Inflammacheck™' device in the diagnosis of COPD.

Participants will be asked to provide an exhaled breath sample for measurement of their EBC H2O2 using 'Inflammacheck™'. The result will be correlated with spirometry (FEV1/ FVC ratio)

DETAILED DESCRIPTION:
A key component of COPD is airway inflammation. Current tools for assessing airway inflammation and oxidative stress, such as fibre-optic bronchoscopy with bronchial wall biopsy and bronchial fluid lavage, are invasive procedures not suitable for routine clinical practice or regular repeat sampling. Sample analysis requires a series of laboratory measurements and results can take over 24 hours to become available.

Non-invasive methods of measuring airway inflammation assess exhaled gases. Fractional exhaled Nitric Oxide (FeNO) measures eosinophilic airway inflammation. However, FeNO does not provide information about neutrophilic airway inflammation, a recognised component of Chronic Obstructive Pulmonary Disease (COPD).

In contrast, measurement of Exhaled Breath Condensate Hydrogen Peroxide (EBC H2O2) is performed during normal tidal breathing, and is well tolerated even in patients with severe airways obstruction and those unable to perform a consistent controlled exhalation. It is also not limited to inflammatory cell specific inflammation. It has the potential to diagnose COPD and to give information about the degree of airway inflammation.

Exhalation Technology Ltd. Have developed a novel, handheld device (Inflammacheck™) which can produce a measurement of EBC H2O2 levels at the patient's side. By detecting EBC H2O2 levels immediately, Inflammacheck™ could tell potentially clinicians and patients the current level of global airway inflammation in a simple, effort independent manner. This could be used by clinicians to diagnose COPD both in hospital and in the community. Previous studies using the 'Inflammacheck™' device have shown that there is a difference in the EBC H2O2 between participants with COPD and those with no underlying lung disease. It has the potential to further measure increased levels of airway inflammation that may indicate an exacerbation of a persons' respiratory disease.

The 'Inflammacheck™' device now requires a study in a clinical setting to validate its use in accurately diagnosing COPD.

The investigators hypothesise that the The 'Inflammacheck™' device will be able to accurately diagnose patients with COPD using EBC H2O2 as compared to the gold standard of Spirometry.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, aged ≥40 years.
* A confirmed, clinician made diagnosis of COPD supported by spirometric evidence of fixed airflow limitation (post-bronchodilator ratio of FEV1/FVC <0.7) recorded at any time.
* OR no known history of lung disease (defined as no current clinical diagnosis of, or be receiving treatment for, a lung disease) and be a current non-smoker. Ex-smokers with a less than 5 pack year history of smoking (cigarettes and cannabis) and who have stopped smoking ≥6 months ago can be included.
* Willing and able to give informed consent for participation in the study.

Exclusion Criteria:

* Existing co-morbidities that may prevent them from performing spirometry (at the discretion of the clinical investigator).
* Known other lung, chest wall, neuromuscular, or cardiac disease (including end-stage disease or cancer) that would confound Inflammacheck™ measurements and spirometry (at the discretion of the clinical investigator).
* Has received treatment for an exacerbation of their COPD within the last 2 weeks.
* In the opinion of the clinical investigator, participant could be put at risk of harm by having to perform any of the study procedures.
* Unable to comprehend the study and provide informed consent e.g. insufficient command of English in the absence of someone to adequately interpret.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: COPD patients and healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 313 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Level of exhaled breath condensate hydrogen peroxide (EBC H2O2) | 1 day study visit
  Respiratory outcome EBC H202 as measured by the inflammacheck sensor
Safety outcome | 1 day study visit
  incidence of adverse events reported during the study procedures
Experience outcome | 1 day study visit
  Rating of ease of use test assessed by Self Completion Questionnaire
Experience outcome | 1 day study visit
  Rating of whether test is acceptable to participant assessed by Self Completion Questionnaire
Experience outcome | 1 day study visit
  Participants' perception of the device assessed by Self Completion Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Portsmouth Hospitals NHS Trust, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No